CLINICAL TRIAL: NCT02856659
Title: Evaluation of N6 Sound Processor in Group of Freedom Users
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CAM5623-FRN6
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Sensory Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study of freedom sound processor users that upgrade to N6 sound processor CP900 series. To test speech understanding in each device and usability of upgrade.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with sensorineural hearing loss
* 12 years of age and older
* Currently using Freedom Sound Processor
* Recipient of a Ci22M or CI24 series implant
* Minimum of 3 months experience with Freedom Sound Processor
* Prior documentation of sentence recognition in noise at a +10 SNR or better
* Native English speaker
* Willingness to participate and comply with requirements of protocol

Exclusion Criteria:

* Unable to complete test metrics
* Unrealistic expectations regarding possible benefits
* Additional handicaps that would prevent or restrict participation in audiological evaluations
* ABI cochlear implant recipient

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children 12 years of age and older.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of N6 Sound Processor in Group of Freedom Users | 3 months of use
  Speech recognition measures in quiet & noise via word and sentence rest and SSiQ questionnaire to compare freedom to upgrade with N6 relative to speech, spatial and quality dimensions and N6 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lori O'Neil, Au.D, Study Director — Cochlear

IPD SHARING:
Plan to Share IPD: Yes